CLINICAL TRIAL: NCT03553082
Title: The Frequency of Airway Complications After LMA Removal in Children: A Comparison of TIVA and Sevoflurane
Brief Title: Airway Complications After LMA in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Jean berezian, Instructor of clinical Anesthesiology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BIO-2017-0276
Record Dates: First submitted 2018-05-08; First posted 2018-06-12 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia Recovery
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthsia (Active Comparator): Patients in this group will receive Propofol 5-6 mg/kg and fentanyl 2 µg/kg for induction of anesthesia and propofol 250-300 µg/kg/min for maintenance.
  Interventions: Drug: Propofol
- Sevoflurane (Active Comparator): Patients in this group will receive sevoflurane 8% and fentanyl 2 µg/kg for induction of anesthesia and sevoflurane 2% for maintenance.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Fentanyl 2 µg/kg for induction of anesthesia and sevoflurane 2% for maintenance
  Arms: Sevoflurane
Drug: Propofol — Propofol 5-6 mg/kg and fentanyl 2 µg/kg for induction of anesthesia and propofol 250-300 µg/kg/min for maintenance
  Arms: Total intravenous anesthsia

SUMMARY:
Background: The removal of Laryngeal Mask Airway (LMA) in children may be associated with respiratory adverse events. The incidence of these adverse events may be influenced by the type of anesthesia maintenance. It is not clear whether Total Intravenous Anesthesia (TIVA) with propofol is associated with a lower incidence of respiratory events upon removal of LMA as compared to maintenance with sevoflurane.

Specific Aim: The primary aim of this study is to compare the prevalence of respiratory adverse events following LMA removal in patient receiving TIVA versus sevoflurane inhalational anesthesia in a pediatric population aged between 6 month and 6 years old. Secondary outcomes include quality of induction, maintenance and emergence from anesthesia between the 2 groups as evidenced by ease of LMA insertion, absence of bucking or movement during the procedure, time to LMA removal, and absence of emergence agitation.

Methods: In this prospective randomized clinical trial, children will be enrolled in one of two groups: Group 1 will receive propofol for induction and maintenance of anesthesia, Group 2 will receive sevoflurane for induction and maintenance of anesthesia. In both groups patients will be mechanically ventilated. At the end of the procedure, LMAs will be removed when patients are fully awake as defined by the return of reflexes, eye opening, and purposeful movements.

Significance: Data comparing the influence of TIVA and sevoflurane on the occurrence of respiratory adverse events after LMA removal are limited. Both techniques are standard of care at our institution. However, as per our clinical observations, we hypothesize that TIVA is superior to sevoflurane. This study will identify the technique that provides optimal anesthetic conditions and improved patient's safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6 months to 6 years old
2. Patients undergoing short duration procedure ( ˂ 2 hours) (such as polysite removal, closed reduction, eye examination, excluding thoracic and abdominal surgery)
3. American Society of Anesthesiologists (ASA): I-III
4. Patients undergoing LMA general anesthesia. (NPO, short procedures, patient without known airway abnormalities).
5. Parental consent

Exclusion Criteria:

1. Age: more than 6 years old and less than 6 months
2. Patients having: Asthma, hyper reactive airway (Acute exacerbation)
3. Patients having recent respiratory tract infection within 2 weeks.
4. Patients with congenital heart disease
5. Patients not eligible for LMA (full stomach, hiatal hernia, known or predicted difficult airway, syndromic patient with facial or airway malformation, patient undergoing major abdominal or thoracic surgery)
6. Patients at high risk of aspiration
7. Anticipated difficult airway
8. Patient with neurologic disorders (children with known neurologic disorders: seizure, mental retardation, cerebral palsy)
9. Difficult LMA insertion (> 3 attempts)

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Respiratory adverse outcomes | 2 hours
  Encountered respiratory adverse outcomes such as cough

SECONDARY OUTCOMES:
Time to emergence | 2 hours
  Emergence time defined as the time from discontinuation of the anesthetic agents until LMA removal.
LMA insertion characteristics | 2 hours
  Number of attempts and time taken to insertion, as well as adverse events encountered during insertion.
Quality of anesthesia | 2 hours
  Lack of movement, bucking, cough
Emergence agitation | 2 hours
  4 points scale: 1: calm, 2: not calm but easily consolable, 3: not easily calmed restless or moderately agitated, 4: combative, disoriented or excited.

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karam C, Zeeni C, Yazbeck-Karam V, Shebbo FM, Khalili A, Abi Raad SG, Beresian J, Aouad MT, Kaddoum R. Respiratory Adverse Events After LMA(R) Mask Removal in Children: A Randomized Trial Comparing Propofol to Sevoflurane. Anesth Analg. 2023 Jan 1;136(1):25-33. doi: 10.1213/ANE.0000000000005945. Epub 2022 Feb 25. PMID 35213484